CLINICAL TRIAL: NCT01881594
Title: Stimulation of Efferent Loop Prior to Ileostomy Closure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Juan Lujan, Section chief. Coloproctology department., Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL-001
Record Dates: First submitted 2013-04-29; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Ileostomy; Complications
Keywords: ileostomy closure,postoperative ileus,stimulation ileostomy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No stimulation (Active Comparator): unstimulated patients prior to surgery,ileostomy closure surgery without prior stimulation of efferent limb.
  Interventions: Procedure: Procedure/Surgery
- Stimulation (Experimental): stimulation of the efferent limb of the ileostomy prior to ileostomy closure.
  Interventions: Procedure: Procedure/Surgery

INTERVENTIONS:
Procedure: Procedure/Surgery — daily stimulation of efferent loop prior to surgery (ileostomy closure)
  Other Names: Stimulation

SUMMARY:
The aim of this study is to compare postoperative ileus between stimulated and unstimulated patients prior to ileostomy closure.

DETAILED DESCRIPTION:
Stimulation was performed ten days prior to the intervention, through the efferent limb of the ileostomy with 500 cc of a thickening substance (saline and nutritional thickener)

ELIGIBILITY:
Inclusion Criteria:

* protective ileostomy after rectal cancer surgery

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
postoperative ileus | within the first days after surgery

REFERENCES:
- [Derived] Abrisqueta J, Abellan I, Lujan J, Hernandez Q, Parrilla P. Stimulation of the efferent limb before ileostomy closure: a randomized clinical trial. Dis Colon Rectum. 2014 Dec;57(12):1391-6. doi: 10.1097/DCR.0000000000000237. PMID 25380005